CLINICAL TRIAL: NCT01954810
Title: Assessment of Antibody Response of a Boosted Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Children Previously Immunized With a Single Dose of JE-CV
Brief Title: Antibody Response of a Boosted Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pope Kosalaraksa, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEC24
Record Dates: First submitted 2013-09-26; First posted 2013-10-07 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Japanese Encephalitis
Keywords: JECV; IMOJEV; Booster response; Children; antibody response; Duration
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Japanese encephaltis chimerix vaccine (No Intervention): This is a single-arm study. Japanese encephalitis chimeric vaccine (JECV) will be administered to all subjects and check for antibody response 4 weeks after vaccination.
  Interventions: Biological: Japanese encephalitis chimeric vaccine (JECV)

INTERVENTIONS:
Biological: Japanese encephalitis chimeric vaccine (JECV) — Japanese encephalitis chimeric vaccine (JECV)will be administered to every children in the study for one dose and check for antibody response 4 weeks after vaccination
  Other Names: IMOJEV

SUMMARY:
This study has aim to describe the immune response to the second dose of Japanese encephalitis chimeric vaccine (JECV) in children previously vaccinated with one dose of JECV 5 years ago.

DETAILED DESCRIPTION:
This is a prospective study to demonstrate the boosting antibody response in children previously vaccinated with one dose of JECV 5 years ago.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who was vaccinated with 1 dose JE-CV in JEC02 and participated in 5 year follow-up in JEC05 trial and finished year 5 of follow-up.
2. Provision of Informed Consent Form signed by at least one parent or other legally acceptable representative.
3. Subject and parent/legally acceptable representative or guardian able to attend all scheduled visits and to comply with all trial procedures
4. In good general health, based on medical history and physical examination

Exclusion Criteria:

1. Participation in another clinical trial investigating a vaccine which need to have vaccination or blood draw within the 4 weeks preceding the trial vaccination except JEC05
2. Planned participation in another clinical trial during the Day0-Day28 period
3. Receipt of live vaccine within 4 weeks preceding the trial vaccination
4. Planned receipt of any vaccine in the 4 weeks following the trial vaccination
5. Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
6. Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
7. Chronic illness or any underlying illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion

Ages: 72 Months to 80 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody titers after JECV vaccination | 28 days
  Neutralizing antibody titers before JECV booster (on D0), and after IMOJEV booster (on D28)

CONTACTS AND LOCATIONS:
Overall Officials: Pope Kosalaraksa, M.D., Principal Investigator — Khon Kaen University
Locations (1):
- Department of Pediatrics, Faculty of Medicine, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand